CLINICAL TRIAL: NCT03127202
Title: Evaluation of Left Ventricular Pacing Vectors Use in Phrenic Nerve Stimulation Management and Left Ventricular Parameters Adjustment
Brief Title: Left Ventricular Pacing Vectors Effectiveness to Narrow Phrenic Nerve Stimulation
Acronym: ORPHEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RTSY01
Record Dates: First submitted 2016-03-02; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac Resynchronization Therapy-Defibrillator (Experimental): Eligible patients were implanted with a Cardiac Resynchronization Therapy -Defibrillator
  Interventions: Device: Cardiac Resynchronization Therapy -Defibrillator (range PARADYM, LivaNova, Clamart, France)

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy -Defibrillator (range PARADYM, LivaNova, Clamart, France) — Patients were implanted with a Cardiac Resynchronization Therapy -Defibrillator (model PARADYM RF SONR CRT-D 9770 or PARADYM RF CRT-D 9750, Sorin) having 3 left ventricular polarities. The choice of the right atrial, right ventricular and bipolar left ventricular leads was left to investigators' discretion.

SUMMARY:
Evaluation of three left ventricular pacing polarities effectiveness to narrow phrenic nerve stimulation.

DETAILED DESCRIPTION:
The primary endpoint of the study aims at demonstrating that the three left ventricular polarities in the Cardiac Resynchronisation Therapy-Defibrillator could bypass phrenic nerve stimulation at least in 90% of implants.

Success was defined as an absence of phrenic nerve stimulation (threshold > 7V) or in case of phrenic nerve stimulation occurrence (threshold < 7V), as the resolution of the phrenic nerve stimulation by reprogramming one of the 3 left ventricular pacing polarities available in the device : left ventricular tip- left ventricular ring (bipolar), left ventricular tip- right ventricular ring (pseudo-bipolar) and left ventricular ring-right ventricular coil.

Any occurrence of phrenic nerve stimulation without resolution by reprogramming was considered as a failure.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for an implantation of a Cardiac Resynchronization Therapy-Defibrillator according to relevant regulations (will be only tolerated primo-implantation and upgrade)
* Patient scheduled for implantation of a Cardiac Resynchronization Therapy-Defibrillator
* Patient has given his informed consent

Exclusion Criteria:

* Any contraindication for Implantable Cardioverter Defibrillator therapy
* Heart transplantation or waiting for heart transplantation
* Implanted with a ventricular assist device (VAD)
* Inability to understand the purpose of the study or to cooperate
* Not available for routine follow-up visits
* Life expectancy less than 12 months
* Age of less than 18 years and et pregnancy
* Under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Phrenic nerve stimulation measurement | The presence of phrenic nerve stimulation will be assessed at implant.
  The presence of phrenic nerve stimulation at 10 Volt, using a pacing system analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Henri BENKEMOUN, Principal Investigator — Clinique Saint Pierre - Perpignan
Locations (12):
- France (12):
  - CH Annecy, Annecy
  - Hopital Henri Mondor, Créteil
  - CH LENS, Lens
  - CH de Bretagne Sud, Lorient
  - Clinique Clairval, Marseille
  - CHP Beauregard, Marseille
  - Clinique Montpellier, Montpellier
  - Polyclinique de Gentilly, Nancy
  - CHU Groupe Hospitalo-universitaire Caremeau, Nîmes
  - Hopital de La Source, Orléans
  - CH St Joseph, Paris
  - Clinique St Pierre, Perpignan

IPD SHARING:
Plan to Share IPD: Undecided